CLINICAL TRIAL: NCT01630447
Title: Identification of Mutations That Lead to Cherubism in Families and Isolated Cases and Studies of Cellular and Molecular Mechanisms
Brief Title: Genetic and Functional Analysis of Cherubism
Acronym: CBM
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Ernst Reichenberger, Assoc. Prof., UConn Health
Other Study IDs: UCHC03-008CBM
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cherubism
Keywords: cherubism; bone; autoinflammatory disorder; osteoblast; osteoclast; mandible; maxilla
MeSH Terms: conditions — Cherubism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood, bone tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this research study is to identify genes and regulatory elements on chromosomes that cause cherubism. Together with the investigators collaborators the investigators also study blood samples and tissue samples from patients to learn about the processes that lead to this disorder. The long-term goal of researchers involved in this study is to find mechanisms to slow down bone resorption in cherubism patients.

DETAILED DESCRIPTION:
Cherubism is a very rare bone disorder where bone gets excessively resorbed only in the jaw bones (mandible and maxilla). The resulting cavities in bone fill up with soft fibrous (fibro-osseous) tissues that can expand and push the bony shells apart. Thus the characteristic facial appearance in patients with progressed cherubism. Bone resorption (cherubism lesions) in this disorder occurs always symmetrically in the mandible, the maxilla or in both. This distinguishes cherubism from similar disorders. As cherubism progresses, the lesions can invade the eye sockets (inferior and/or lateral orbital walls) and displace the eye balls and push down the eyelids. As a result the sclera (white of the eye) below the iris becomes visible and patients have an upward gazing appearance (cherubic look) which gave the name to this fibro-proliferative bone disorder.

Cherubism typically appears between ages of 2-7 years. It is often diagnosed during dental evaluations. At early stages cherubism is accompanied by lymph node swelling. Proliferation of the fibro-osseous tissue typically stops after puberty and in many the soft tissue in the cherubic bone cavities are replaced by new bone.

For this study we will:

* Send out study participation kits and consent by phone
* Collect a saliva sample from eligible individuals
* Obtain information regarding cherubism
* Document disorder with photos and doctor's letters
* If patients undergo surgery for cherubism we ask to obtain some bone tissue that would otherwise be discarded
* Isolate DNA from the saliva sample
* Perform genetic analyses of the DNA with the most up-to-date methods available to identify genetic variations
* Study in the laboratory why the genetic variations cause the disorder

ELIGIBILITY:
Inclusion Criteria:

* cherubism; unaffected individuals only if part of a participating cherubism family

Exclusion Criteria:

* no cherubism unaffected individuals only as part of a participating cherubism family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with clinically diagnosed cherubism
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-04; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic elements | at time of identification
  The goal is to identify relevant genes or genetic elements that cause the disease or contribute to the disease progression and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst J Reichenberger, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Levaot N, Voytyuk O, Dimitriou I, Sircoulomb F, Chandrakumar A, Deckert M, Krzyzanowski PM, Scotter A, Gu S, Janmohamed S, Cong F, Simoncic PD, Ueki Y, La Rose J, Rottapel R. Loss of Tankyrase-mediated destruction of 3BP2 is the underlying pathogenic mechanism of cherubism. Cell. 2011 Dec 9;147(6):1324-39. doi: 10.1016/j.cell.2011.10.045. PMID 22153076
- [Result] Ueki Y, Tiziani V, Santanna C, Fukai N, Maulik C, Garfinkle J, Ninomiya C, doAmaral C, Peters H, Habal M, Rhee-Morris L, Doss JB, Kreiborg S, Olsen BR, Reichenberger E. Mutations in the gene encoding c-Abl-binding protein SH3BP2 cause cherubism. Nat Genet. 2001 Jun;28(2):125-6. doi: 10.1038/88832. PMID 11381256
- [Result] Gilbert G, Defillo M, Delcan JL, David P. [Results of anastomoses in the tetralogy of Fallot]. Union Med Can. 1966 Dec;95(12):1377-84. No abstract available. French. PMID 5996221
- [Result] Ueki Y, Lin CY, Senoo M, Ebihara T, Agata N, Onji M, Saheki Y, Kawai T, Mukherjee PM, Reichenberger E, Olsen BR. Increased myeloid cell responses to M-CSF and RANKL cause bone loss and inflammation in SH3BP2 "cherubism" mice. Cell. 2007 Jan 12;128(1):71-83. doi: 10.1016/j.cell.2006.10.047. PMID 17218256
- [Result] Wang CJ, Chen IP, Koczon-Jaremko B, Boskey AL, Ueki Y, Kuhn L, Reichenberger EJ. Pro416Arg cherubism mutation in Sh3bp2 knock-in mice affects osteoblasts and alters bone mineral and matrix properties. Bone. 2010 May;46(5):1306-15. doi: 10.1016/j.bone.2010.01.380. Epub 2010 Feb 1. PMID 20117257
- [Result] Levaot N, Simoncic PD, Dimitriou ID, Scotter A, La Rose J, Ng AH, Willett TL, Wang CJ, Janmohamed S, Grynpas M, Reichenberger E, Rottapel R. 3BP2-deficient mice are osteoporotic with impaired osteoblast and osteoclast functions. J Clin Invest. 2011 Aug;121(8):3244-57. doi: 10.1172/JCI45843. Epub 2011 Jul 18. PMID 21765218
- [Result] Reichenberger EJ, Levine MA, Olsen BR, Papadaki ME, Lietman SA. The role of SH3BP2 in the pathophysiology of cherubism. Orphanet J Rare Dis. 2012 May 24;7 Suppl 1(Suppl 1):S5. doi: 10.1186/1750-1172-7-S1-S5. Epub 2012 May 24. PMID 22640988
- [Result] Papadaki ME, Lietman SA, Levine MA, Olsen BR, Kaban LB, Reichenberger EJ. Cherubism: best clinical practice. Orphanet J Rare Dis. 2012 May 24;7 Suppl 1(Suppl 1):S6. doi: 10.1186/1750-1172-7-S1-S6. Epub 2012 May 24. PMID 22640403
- [Result] Yoshimoto T, Hayashi T, Kondo T, Kittaka M, Reichenberger EJ, Ueki Y. Second-Generation SYK Inhibitor Entospletinib Ameliorates Fully Established Inflammation and Bone Destruction in the Cherubism Mouse Model. J Bone Miner Res. 2018 Aug;33(8):1513-1519. doi: 10.1002/jbmr.3449. Epub 2018 May 22. PMID 29669173
- [Result] Yoshitaka T, Mukai T, Kittaka M, Alford LM, Masrani S, Ishida S, Yamaguchi K, Yamada M, Mizuno N, Olsen BR, Reichenberger EJ, Ueki Y. Enhanced TLR-MYD88 signaling stimulates autoinflammation in SH3BP2 cherubism mice and defines the etiology of cherubism. Cell Rep. 2014 Sep 25;8(6):1752-1766. doi: 10.1016/j.celrep.2014.08.023. Epub 2014 Sep 15. PMID 25220465
- [Result] Mione MC, Dhital KK, Amenta F, Burnstock G. An increase in the expression of neuropeptidergic vasodilator, but not vasoconstrictor, cerebrovascular nerves in aging rats. Brain Res. 1988 Sep 13;460(1):103-13. doi: 10.1016/0006-8993(88)91210-3. PMID 3265349
- [Result] Kittaka M, Yoshimoto T, Schlosser C, Kajiya M, Kurihara H, Reichenberger EJ, Ueki Y. Microbe-Dependent Exacerbated Alveolar Bone Destruction in Heterozygous Cherubism Mice. JBMR Plus. 2020 Apr 14;4(6):e10352. doi: 10.1002/jbm4.10352. eCollection 2020 Jun. PMID 32537546
- [Result] Fujii Y, Monteiro N, Sah SK, Javaheri H, Ueki Y, Fan Z, Reichenberger EJ, Chen IP. Tlr2/4-Mediated Hyperinflammation Promotes Cherubism-Like Jawbone Expansion in Sh3bp2 (P416R) Knockin Mice. JBMR Plus. 2021 Oct 30;6(1):e10562. doi: 10.1002/jbm4.10562. eCollection 2022 Jan. PMID 35079675
- See also: Description of lab research and patient recruitment procedures — https://health.uconn.edu/reichenberger-lab/